CLINICAL TRIAL: NCT04831749
Title: Cross-cultural Translation and Validation of the Quebec Back Pain Disability Scale Into Local Languages of Pakistan.
Brief Title: Translation of Quebec Back Pain Disability Scale Into Local Languages of Pakistan.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00932 Sana Hanif
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Quebec Back Pain Disability Scale; Tool Translation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to translate the Quebec Back Pain Disability Scale into Pashto, Punjabi, Sindhi and Balochi languages. Along with validation of the translated versions by evaluating their validity and reliability in the people of Pakistan, speaking respective languages and suffering from low back pain. No such study has been previously conducted in the Pakistan region which translates the scale and follows the proper cross-culture adaptation.

DETAILED DESCRIPTION:
The Quebec Back Pain Disability Scale is a first-hand measure of functional disability for patients with back pain. It distinguishes itself from other published scales as it has an approach that deals with the concepts of disability and its assessment. Its major aim is to be a responsive measure of functional disability in back pain. Quebec back pain disability Questionnaire has unique strong characteristics that are quite feasibly used and have good identification properties regarding Low Back Pain. There is extensive usage, applicability, and validity of QBPDS in research and clinical practice. Along with these factors the capability of the QBPDS to identify significant fluctuations in patient's condition, makes its use evidently advocated.

Quebec Pain disability scale, originally a French scale has been translated and validated into a few languages before. Previous studies have shown that the translation of the scale would end up giving a standard measure to be utilized in clinical practices and research studies while sanctioning clinicians and specialists to share information and to study effects of treatments in low back pain patients. Along with helping in appraisals of outcomes amongst various populations. So, to gather the best outcomes of this questionnaire in Pakistan region it is imperative to translate it into Pashto, Punjabi, Sindhi and Balochi hence the local languages.

ELIGIBILITY:
Inclusion Criteria:

* Patients both male and female having age group equal or >18,
* should be able to read the questionnaire that is in their native language(Punjabi, Sindhi, Balochi and Pashto) and
* diagnosed with nonspecific low back pain for more than 3 months.

Exclusion Criteria:

* Any serious conditions like neurological conditions which would not allow the patient to fill the questionnaire independently,
* any infection, tumor, spinal surgery, cognitive impairments, or any other rheumatologic disease would be excluded.
* Any issues in understanding or expressing the native language (Punjabi, Pashto, Balochi or Sindhi) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To meet inclusion criteria participants diagnosed with low back pain, clinically stable, and able to read the local language version of QBPDS. Then patient response will be checked on the translated versions
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Cross-Cultural Translation of Quebec Back Pain Disability Scale into the local languages (Punjabi, Pashto, Sindhi, Balochi) | 6 months
  The Quebec Back Pain Disability Scale is a first-hand measure of functional disability for patients with back pain. The scale has 20 items, representing six empirically derived categories of activities affected by back pain. It is an self-administered tool targeted on the population with Low back pain. It distinguishes itself from other published scales as it has an approach that deals with the concepts of disability and its assessment. Its translation is to be done in local languages of Pakistan through a rigorous and approved process

SECONDARY OUTCOMES:
reliability and validity of translated versions | 6 months
  To determine reliability and validity of cross-culturally adapted and the translated QBPDS versions in patients with low back pain of respective languages۔ Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two or more interval between different visits of the patient and validity is how accurate the results are. Thus these both are to measured through various parameters to validate the translated versions as appropriate and applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Ali Muhammad Memorial, Multan, Punajb, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN checklist for assessing the methodological quality of studies on measurement properties of health status measurement instruments: an international Delphi study. Qual Life Res. 2010 May;19(4):539-49. doi: 10.1007/s11136-010-9606-8. Epub 2010 Feb 19. PMID 20169472
- [Background] Zaidi S, Verma S, Moiz JA, Hussain ME. Transcultural adaptation and validation of Hindi version of Quebec Back Pain Disability Scale. Disabil Rehabil. 2018 Dec;40(24):2938-2945. doi: 10.1080/09638288.2017.1362596. Epub 2017 Aug 7. PMID 28783980
- [Background] Monticone M, Frigau L, Mola F, Rocca B, Franchignoni F, Simone Vullo S, Foti C, Chiarotto A. The Italian version of the Quebec Back Pain Disability Scale: cross-cultural adaptation, reliability and validity in patients with chronic low back pain. Eur Spine J. 2020 Mar;29(3):530-539. doi: 10.1007/s00586-019-06153-4. Epub 2019 Sep 26. PMID 31559506
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Hafeez A. Urdu version of the neck disability index: a reliability and validity study. BMC Musculoskelet Disord. 2017 Apr 8;18(1):149. doi: 10.1186/s12891-017-1469-5. PMID 28388888